CLINICAL TRIAL: NCT05076656
Title: Epigenetic and Microbiota Modifications in the Genesis of Adipose Tissue Dysfunction
Brief Title: Epigenetic and Microbiota Modifications
Acronym: EPI-MICROBIO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EPIGEN-MICROBIOTA
Record Dates: First submitted 2021-09-15; First posted 2021-10-13 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2021-07

CONDITIONS: Diabetes type2; Obesity
Keywords: Diabetes type2; FMT; Probiotics; Microbiota
MeSH Terms: conditions — Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics arm (Experimental): Individuals who receive a probiotics pill daily: Lactobacillus fermentum D3 (PCT/EP 2012058214)
  Interventions: Dietary Supplement: Lactobacillus fermentum D3
- FMT arm (Experimental): Individuals who receive a FMT in the form of pills with fecal material from a healthy donor.
  Interventions: Biological: Fecal microbiota transplant (FMT)
- Control arm (Placebo Comparator): Individuals who receive a probiotics pill daily of placebo (milk powder)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus fermentum D3 — Lactobacillus fermentum D3 in a white, gelatin capsule (orally), with lyophilized L. fermentum D3 without preservatives, sugars, or additives.
  Other Names: PCT/EP 2012058214
  Arms: Probiotics arm
Biological: Fecal microbiota transplant (FMT) — Fecal microbiota transplant (FMT) in a green, gelatin capsule (orally), with lyophilized fecal material.
  Arms: FMT arm
Drug: Placebo — Placebo in a white, gelatin capsule (orally), with powder milk
  Arms: Control arm

SUMMARY:
In order to investigate how gut microbiota interventions are able to change gut microbiota population and impact insulin resistance, 30 type2 diabetes volunteers with obesity will be randomized to one of the three treatment groups: 1) probiotics arm, who will take a Lactobacillus fermentum D3 in pills daily; 2) FMT arm, who will take a lyophilized fecal microbiota transplant in pills; and 3) control group, who will take placebo pills. After 3 months, insulin resistance, glucose metabolism parameters, and gut microbiota variation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Type2 diabetes in treatment with metformin
* 30 kg/m2≤IMC≤40 kg/m2
* 30-70 years old
* HOMA-IR >6
* Informed consent

Exclusion Criteria:

* psychopathologic alterations that do not permit the adherence to the trial.
* Diabetes medication different from metformin.
* History of cholecystectomy.
* Use of Probiotics, and/or antibiotics in the last 3 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in HOMA-IR | Baseline, 12 weeks
  Homeostasis Model Assessment of fasting Insulin Resistance (HOMA-IR: glucose (mmol/l( x insulin (pmol/l)/22.5)

SECONDARY OUTCOMES:
Changes in gut microbiota | Baseline, 12 weeks
  Change from baseline in 16S rRNA amplicons after 3 months
Changes in glucose metabolism | Baseline, 12 weeks
  Change from baseline in oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Tinahones, MD, PhD, Principal Investigator — Instituto de Investigacion Biomedica de Malaga
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain